CLINICAL TRIAL: NCT00767507
Title: BRIDGE: Maintenance of Platelet inihiBition With cangRelor After dIscontinuation of ThienopyriDines in Patients Undergoing surGEry
Brief Title: Maintenance of Platelet Inhibition With Cangrelor
Acronym: Bridge
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TMC-CAN-08-02
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Results first posted 2014-04-04 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-02

CONDITIONS: Acute Coronary Syndrome (ACS)
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — cangrelor

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cangrelor (Experimental): Cangrelor was administered as a continuous IV infusion of 0.75µg/kg/min for a minimum of 48 hours and a maximum of 7 days.
  Interventions: Drug: cangrelor
- Placebo (Placebo Comparator): A placebo infusion was administered as a continuous IV infusion of 0.75µg/kg/min for a minimum of 48 hours and a maximum of 7 days, to maintain the blind.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: cangrelor
  Arms: Cangrelor
Other: Placebo — Placebo IV infusion administered in the same fashion as the active study drug in order to maintain the blind in the study.
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate that patients receiving cangrelor infusion before coronary artery bypass grafting have an acceptable safety profile and can undergo surgery without excessive bleeding peri-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* 18 Years of Age
* Non emergent coronary bypass graft surgery
* Received a thienopyridine within 48 hours prior to enrollment

Exclusion Criteria:

* Confirmed or suspected pregnancy
* Cerebrovascular accident within one yar
* Intracranial neoplasm
* History of bleeding diathesis
* Thrombocytopenia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2008-10; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Topol, MD, Principal Investigator — Scripps
Locations (1):
- Scripps Clinic / Scripps Green Hospital, La Jolla, California, United States

REFERENCES:
- [Derived] Angiolillo DJ, Firstenberg MS, Price MJ, Tummala PE, Hutyra M, Welsby IJ, Voeltz MD, Chandna H, Ramaiah C, Brtko M, Cannon L, Dyke C, Liu T, Montalescot G, Manoukian SV, Prats J, Topol EJ; BRIDGE Investigators. Bridging antiplatelet therapy with cangrelor in patients undergoing cardiac surgery: a randomized controlled trial. JAMA. 2012 Jan 18;307(3):265-74. doi: 10.1001/jama.2011.2002. PMID 22253393

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients with acute coronary syndrome (ACS) or who had previously received stents, who were required to discontinue maintenance oral P2Y12 therapy before cardiac surgery. Patients who had discontinued oral therapy within the previous 72 hours were eligible. Patients were hospitalized during the enrollment period.
Pre-assignment Details: Stage I was an open-label, dose-finding stage to identify the dose of cangrelor that achieved a level of antiplatelet effect after discontinuation of oral P2Y12 therapy equivalent to the previous oral P2Y12 maintenance therapy. These patients were not enrolled in Stage II.
  Stage II was randomized, double-blind, placebo-controlled.
Groups:
- Stage I, Cohort I - 0.5 mcg/kg/Min Cangrelor: Patients who received cangrelor as a continuous IV infusion of 0.5 mcg/kg/min for a minimum of 48 hours and a maximum of 7 days.
- Stage I, Cohort II - 0.75 mcg/kg/Min Cangrelor; Stage II - Cangrelor Arm (0.75 mcg/kg/Min ): Patients who received cangrelor as a continuous IV infusion of 0.75 mcg/kg/min for a minimum of 48 hours and a maximum of 7 days.
- Stage II - Placebo Arm: Patients who received matching placebo as a continuous IV infusion of 0.75 mcg/kg/min for a minimum of 48 hours and a maximum of 7 days.
Period: Overall Study
Arm/Group | Stage I, Cohort I - 0.5 mcg/kg/Min Cangrelor | Stage I, Cohort II - 0.75 mcg/kg/Min Cangrelor | Stage II - Cangrelor Arm (0.75 mcg/kg/Min ) | Stage II - Placebo Arm
Started | 5 | 6 | 106 | 104
Completed | 5 | 6 | 106 | 101
Not Completed | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: This is the Safety Population: Includs both Stage I and Stage II patients who received any study drug and were classified according to the actual treatment received. Stage I (open-label) patients were analyzed based on the dose they received; Stage II (randomized) patients were analyzed based on the actual treatment, cangrelor or placebo, received.
Groups:
- Stage II Cangrelor Arm (0.75 mcg/kg/Min): Patients who received cangrelor as a continuous IV infusion of 0.75 mcg/kg/min for a minimum of 48 hours and a maximum of 7 days.
- Stage II Placebo Arm: Patients who received matching placebo as a continuous IV infusion of 0.75 mcg/kg/min for a minimum of 48 hours and a maximum of 7 days.
- Total: Total of all reporting groups
Arm/Group | Stage I, Cohort I - 0.5 mcg/kg/Min Cangrelor | Stage I, Cohort II - 0.75 mcg/kg/Min Cangrelor | Stage II Cangrelor Arm (0.75 mcg/kg/Min) | Stage II Placebo Arm | Total
Number analyzed (Participants) | 5 | 6 | 106 | 101 | 218
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 52 | 59 | 117
  >=65 years | 2 | 3 | 54 | 42 | 101
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 26 | 27 | 55
  Male | 5 | 4 | 80 | 74 | 163
Region of Enrollment [Number; unit: participants] — This population in Region of Enrollment, represents the total number of subjects enrolled/randomized, and does not exclude any patients. Therefore there are more patients represented here versus in the Safety Population.
  participants
    United States | 5 | 6 | 66 | 59 | 136
    Netherlands | 0 | 0 | 5 | 6 | 11
    Czech Republic | 0 | 0 | 26 | 29 | 55
    United Kingdom | 0 | 0 | 8 | 4 | 12
    Austria | 0 | 0 | 1 | 6 | 7

OUTCOME MEASURES:

1. Primary Outcome: Stage I: Percentage of Patient Samples That Maintained Platelet Inhibition Levels of Greater Than or Equal to 60% as Reported by the VerifyNow P2Y12 Point of Care Assay.
Description: Endpoint was selected as an approximation of the antiplatelet effect expected to be maintained if oral P2Y12 inhibitors had not been discontinued (60% inhibition of platelets).
Time Frame: During study drug infusion up to 1-6 hours prior to surgery
Measure: Number; unit: percentage of samples
Units Other Than Participants: samples
Groups:
- Stage I, Cohort I - Cangrelor 0.5 mcg/kg/Min: Patients who received cangrelor as a continuous IV infusion of 0.5 mcg/kg/min for a minimum of 48 hours and a maximum of 7 days.
- Stage I, Cohort II - Cangrelor 0.75 mcg/kg/Min: Patients who received cangrelor as a continuous IV infusion of 0.75 mcg/kg/min for a minimum of 48 hours and a maximum of 7 days.
Arm/Group | Stage I, Cohort I - Cangrelor 0.5 mcg/kg/Min | Stage I, Cohort II - Cangrelor 0.75 mcg/kg/Min
Number analyzed (Participants) | 5 | 6
Number analyzed (samples) | 17 | 18
percentage of samples | 76.5 | 94.4

2. Primary Outcome: Stage II: The Percentage of Patients That Maintained Platelet Reaction Units (PRU) < 240, as Determined by the VerifyNow P2Y12 Point of Care Assay, Measured During Study Drug Infusion Pre-surgery.
Description: This endpoint was selected as it is considered by consensus of the Working Group on Platelet Reactivity to be the threshold for the level of platelet inhibition required to maintain a low risk of coronary thrombosis and cardiac ischemic events.
  Patients had multiple samples and all "on-infusion" samples had to be <240 PRU to meet the endpoint.
Time Frame: During study drug infusion up to 1-6 hours prior to surgery
Population: Based on available data from ITT population; ITT population (Cangrelor N = 93) / (Placebo N = 90).
  Valid PRU results were not available during the infusion period for 15 patients (9 cangrelor and 6 placebo).
Measure: Number; unit: Percent of patients
Groups:
- Stage II - Cangrelor Arm (0.75 mcg/kg/Min): Patients who received cangrelor as a continuous IV infusion of 0.75 mcg/kg/min for a minimum of 48 hours and a maximum of 7 days.
- Stage II - Placebo Arm: Patients who received m as a matching placebo as a continuous IV infusion of 0.75 mcg/kg/min for a minimum of 48 hours and a maximum of 7 days.
Arm/Group | Stage II - Cangrelor Arm (0.75 mcg/kg/Min) | Stage II - Placebo Arm
Number analyzed (Participants) | 84 | 84
Percent of patients | 98.8 | 19.0

3. Secondary Outcome: Stage II: Analysis of Platelet Reactivity (ITT Population) / Patients With Platelet Reactivity < 240 PRU
Description: This endpoint analyzed the percent of patients with platelet reactivity < 240 PRU at the following timepoints:
  * Baseline - Prior to study drug infusion (washout period from oral P2Y12 inhibition)
  * Last sample during infusion
  * Following discontinuation of study drug infusion
Time Frame: baseline until just prior to surgery (post infusion)
Measure: Number; unit: percent of patients
Arm/Group | Stage II - Cangrelor Arm (0.75 mcg/kg/Min) | Stage II - Placebo Arm
Number analyzed (Participants) | 93 | 90
percent of patients
  Prior to study drug infusion (washout period) | 62.4 | 52.3
  Last sample during infusion | 98.8 | 31.0
  Following discontinuation of study drug infusion | 26.9 | 20.0

4. Secondary Outcome: Incidence of Excessive Coronary Artery Bypass Graft (CABG)-Related Bleeding
Description: Defined as the occurrence of surgical re-exploration, 24-hour chest tube output of >1.5 liters (L), and/or packed red blood cell transfusions > 4 units
Time Frame: Randomization through Hospital discharge
Population: This analysis included only those patients who proceeded to have a CABG surgery as required per the protocol. The patients who did not have a CABG surgery were excluded from the denominator.
Measure: Number; unit: Patients
Arm/Group | Stage II - Cangrelor Arm (0.75 mcg/kg/Min) | Stage II - Placebo Arm | Stage I, Cohort I - Cangrelor 0.5 mcg/kg/Min | Stage I, Cohort II - Cangrelor 0.75 mcg/kg/Min
Number analyzed (Participants) | 102 | 96 | 5 | 6
Patients | 12 | 10 | 0 | 1

5. Secondary Outcome: Non-CABG (Preoperative) Bleeding - Protocol-defined GUSTO Severe/Life-threatening, Moderate and Mild
Time Frame: Randomization until start of CABG surgery
Population: as for outcome 4
Measure: Number; unit: participants
Groups:
- Stage II - Cangrelor (0.75 mcg/kg/Min); Stage I, Cohort II - Cangrelor 0.75 mcg/kg/Min: Patients who received cangrelor as a continuous IV infusion of 0.75 mcg/kg/min for a minimum of 48 hours and a maximum of 7 days.
- Stage I, Cohort 1 - Cangrelor 0.5 mcg/kg/Min: Patients who received cangrelor as a continuous IV infusion of 0.5 mcg/kg/min for a minimum of 48 hours and a maximum of 7 days.
Arm/Group | Stage II - Cangrelor (0.75 mcg/kg/Min) | Stage II - Placebo Arm | Stage I, Cohort 1 - Cangrelor 0.5 mcg/kg/Min | Stage I, Cohort II - Cangrelor 0.75 mcg/kg/Min
Number analyzed (Participants) | 102 | 96 | 5 | 6
participants
  GUSTO severe/life threatening | 2 | 1 | 0 | 0
  GUSTO moderate | 10 | 4 | 0 | 2
  GUSTO mild | 8 | 5 | 1 | 1

6. Secondary Outcome: Patients With Blood Product Transfusions up to 7 Days After Surgery or Discharge, Whichever Was Sooner
Time Frame: Through 7 days or hospital discharge, whichever was sooner
Measure: Number; unit: patients
Groups:
- Stage I, Cohort 1 - Cangrelor (0.5 mcg/kg/Min): Patients who received cangrelor as a continuous IV infusion of 0.5 mcg/kg/min for a minimum of 48 hours and a maximum of 7 days.
- Stage I - Cohort II - Cangrelor 0.75 mcg/kg/Min: Patients who received cangrelor as a continuous IV infusion of 0.75 mcg/kg/min for a minimum of 48 hours and a maximum of 7 days.
Arm/Group | Stage II - Cangrelor Arm (0.75 mcg/kg/Min) | Stage II - Placebo Arm | Stage I, Cohort 1 - Cangrelor (0.5 mcg/kg/Min) | Stage I - Cohort II - Cangrelor 0.75 mcg/kg/Min
Number analyzed (Participants) | 106 | 101 | 5 | 6
patients | 34 | 35 | 1 | 4

ADVERSE EVENTS:
Arm/Group | Stage I, Cohort I - Cangrelor 0.5 mcg/kg/Min | Stage I, Cohort II - Cangrelor 0.75 mcg/kg/Min | Stage II - Cangrelor Arm (0.75 mcg/kg/Min) | Stage II - Placebo Arm
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 11/106 | 9/101
Other Adverse Events (participants affected / at risk) | 3/5 | 5/6 | 27/106 | 23/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage I, Cohort I - Cangrelor 0.5 mcg/kg/Min (N=5) | Stage I, Cohort II - Cangrelor 0.75 mcg/kg/Min (N=6) | Stage II - Cangrelor Arm (0.75 mcg/kg/Min) (N=106) | Stage II - Placebo Arm (N=101)
angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
cardiac arrest (Cardiac disorders) | 0 | 0 | 3 | 1
cardiac asthma (Cardiac disorders) | 0 | 0 | 0 | 1
cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 2
cardiogenic shock (Cardiac disorders) | 0 | 0 | 4 | 1
cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 0 | 1
coronary artery thrombosis (Cardiac disorders) | 0 | 0 | 1 | 0
papillary muscle rupture (Cardiac disorders) | 0 | 0 | 1 | 0
ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
chest pain (General disorders) | 0 | 0 | 1 | 0
multi-organ failure (General disorders) | 0 | 0 | 0 | 1
systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1 | 0
abdominal sepsis (Infections and infestations) | 0 | 0 | 0 | 1
beta haemolytic streptococcal infection (Infections and infestations) | 0 | 0 | 1 | 0
gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 0 | 1
mediastinitis (Infections and infestations) | 0 | 0 | 1 | 0
vasoplegia syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0
bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
arterial thrombosis limb (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stage I, Cohort I - Cangrelor 0.5 mcg/kg/Min (N=5) | Stage I, Cohort II - Cangrelor 0.75 mcg/kg/Min (N=6) | Stage II - Cangrelor Arm (0.75 mcg/kg/Min) (N=106) | Stage II - Placebo Arm (N=101)
angina pectoris (Cardiac disorders) | 0 | 1 | 3 | 0
overdose (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 5
arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0
atrial fibrillation (Cardiac disorders) | 0 | 1 | 1 | 5
pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 2
tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0
ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
nausea (Gastrointestinal disorders) | 0 | 1 | 10 | 3
toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
discomfort (General disorders) | 0 | 1 | 1 | 0
pyrexia (General disorders) | 1 | 0 | 1 | 3
anemia postoperative (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
incision site pain (Injury, poisoning and procedural complications) | 1 | 1 | 11 | 8
procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
white blood cell count increased (Investigations) | 0 | 1 | 0 | 0
fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 3 | 0
back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 3
lethargy (Nervous system disorders) | 0 | 1 | 0 | 1
metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
agitation (Psychiatric disorders) | 0 | 1 | 3 | 1
confusional state (Psychiatric disorders) | 0 | 1 | 1 | 1
disorientation (Psychiatric disorders) | 0 | 1 | 2 | 0
restlessness (Psychiatric disorders) | 0 | 1 | 3 | 0
azotaemia (Renal and urinary disorders) | 0 | 2 | 0 | 0
bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
constipation (Gastrointestinal disorders) | 0 | 0 | 7 | 2
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6 | 1
anxiety (Psychiatric disorders) | 0 | 0 | 7 | 2
insomnia (Psychiatric disorders) | 0 | 0 | 6 | 1
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, PI communications regarding trial results are prohibited until after the communication and publication of the multi-center results by Sponsor, but no more than 12 months after conclusion of the trial at all sites.

PI must submit results communications to sponsor for review at least 60 days prior to submission for publication and Sponsor may embargo such communications for a period that is less than or equal to 150 days solely to seek appropriate patent protection.